CLINICAL TRIAL: NCT01214733
Title: An Open Label Study of the Safety During Treatment With Tocilizumab (TCZ), in Combination With Disease Modifying Anti-rheumatic Drugs (DMARDs), in Patients With Moderate to Severe Rheumatoid Arthritis
Brief Title: A Study of RoActemra/Actemra (Tocilizumab) Plus DMARDs in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25321
Record Dates: First submitted 2010-10-04; First posted 2010-10-05 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] — 8 mg/kg intravenously every 4 weeks in combination with allowed DMARDs

SUMMARY:
This open-label study will evaluate the long-term safety and efficacy of RoActemra/Actemra (tocilizumab) in combination with disease modifying anti-rheumatic drugs (DMARDs) in patients with moderate to severe rheumatoid arthritis. Patients who successfully completed studies WA17823 and WA18696 in South Africa are eligible to participate in this study. Patients will be allowed DMARDs according to the treatment they received in the previous studies. Patients will receive 8 mg/kg RoActemra/Actemra intravenously every 4 weeks. The anticipated time on study treatment is 104 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/=18 years of age
* Moderate to severe rheumatoid arthritis of more than 6 months duration upon entering the study
* Patients successfully completed studies WA17823 and WA18696 in South Africa
* Body weight <150 kg

Exclusion Criteria:

* Patients who have withdrawn from studies WA17823 and WA18696 are not eligible to participate in this study Treatment with any investigational agent since last administration of study drug in studies WA17823 and WA18696
* Previous treatment with any cell depleting therapies
* Treatment with intravenous gamma globulin, plasmapheresis or Prosorba(TM) column since the last administration of study drug in studies WA17823 and WA18696

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Safety (incidence of adverse events) | 104 weeks
Safety (laboratory assessments e.g. hematology) | 104 weeks

SECONDARY OUTCOMES:
Efficacy: Change in Disease Activity Score (DAS28) | 104 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- South Africa (2):
  - Cape Town
  - Diepkloof